CLINICAL TRIAL: NCT01558362
Title: A Phase 1 Study of Safety, Tolerance, Pharmacokinetics and Nuclear Medicine Imaging of 123I-CMICE-013 Administered Intravenously in Healthy Adult Volunteers
Brief Title: A Study of 123I-CMICE-013 Radiopharmaceutical in Healthy Volunteers
Acronym: CMICE
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 20120080-01H
Record Dates: First submitted 2012-03-07; First posted 2012-03-20 (Estimated); Results first posted 2025-03-26 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-01

CONDITIONS: Coronary Artery Disease
Keywords: myocardial perfusion imaging; single photon emission tomography; Coronary artery disease; gamma camera imaging; Phase 1 clinical trial; cyclotron
MeSH Terms: conditions — Coronary Artery Disease | interventions — CMICE-013

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 123I-CMICE-013 (Experimental): Administration and analysis of alternative MPI radiotracer
  Interventions: Drug: 123I-CMICE-013

INTERVENTIONS:
Drug: 123I-CMICE-013 — 2 intravenous doses of drug will be given one week apart. Doses will be equivalent to 1 rest dose and 1 stress dose. Serial nuclear imaging will follow dose injections. All volunteers had a rest dose first followed by a stress dose.

SUMMARY:
The need exists for alternatives to 99mTc based perfusion radiotracers for cardiac patient management. An alternative radiotracer, I123-CMICE-013, has been developed at the Canadian Molecular Imaging Center of Excellence (C-MICE) at the University of Ottawa Heart Institute. Initial testing results in rats and pigs suggest that in addition to being a cyclotron-produced alternative to 99mTc tracers, I-123-CMICE-013 may be a superior tracer for measuring myocardial perfusion.This Phase 1 study will study the safety and tolerability, biodistribution, pharmacokinetics and radiation dosimetry, and distribution and localization of I123-CMICE-013in healthy adult volunteers.

DETAILED DESCRIPTION:
Single photon emission computed tomography (SPECT) myocardial perfusion imaging (MPI) is an established, cost effective tool for the risk stratification and management of patients suspected or known to have coronary artery disease (CAD)Myocardial perfusion imaging is significantly affected by interruptions in the supply of 99mMo, the parent isotope of 99mTc used for the majority of MPI. An alternative radiotracer, I123-CMICE-013,developed at the Canadian Molecular Imaging Center of Excellence (C-MICE) at the University of Ottawa Heart Institute, has completed pre-clinical trial testing and is ready for Phase 1 human trials.

This Phase I study will be a single centre, open label study. Subjects will receive 2 doses of study drug. One rest dose and one stress dose will be administered on separate days, one week apart. Subjects will undergo a standard clinical exercise stress protocol for the stress dose. Gamma camera imaging following each administration will be done over 2 days.

Biodistribution, pharmacokinetics, dosimetry and safety variables will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 65 years
2. No significant medical history
3. Normal physical exam
4. BMI ≤ 30 kg/m2
5. No current use of prescription medication
6. No clinically significant abnormalities in baseline laboratory work
7. No clinically significant abnormalities in baseline 12 lead electrocardiogram
8. Female subjects must be post-menopausal, surgically sterilized or have negative urine beta human chorionic gonadotropin pregnancy test at initial screening

Exclusion Criteria:

1. Pregnancy
2. Known hypersensitivity to the investigational drug or any of its components
3. Claustrophobia or inability to lie still in a supine position
4. Unwillingness to provide informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-04; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Terrence D Ruddy, MD, Principal Investigator — Ottawa Heart Institute Research Corporation
Locations (1):
- University of Ottawa Heart Institute, Ottawa, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 12 healthy normal volunteers will be recruited to complete the study.
Groups:
- 123I-CMICE-013: Administration and analysis of alternative MPI radiotracer
  123I-CMICE-013: 2 identical doses of intravenous drug will be given one week apart. Rest imaging will follow the initial dose. Exercise treadmill stress testing will follow the second dose. Serial nuclear imaging will follow dose injections.
Period: Overall Study
Arm/Group | 123I-CMICE-013
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- 123I-CMICE-013: Administration and analysis of alternative MPI radiotracer
  123I-CMICE-013: 2 intravenous doses of drug will be given one week apart. Doses will be equivalent to 1 rest dose and 1 stress dose. Serial nuclear imaging will follow dose injections.
Arm/Group | 123I-CMICE-013
Number analyzed (Participants) | 12
Age, Continuous [Mean (Full Range); unit: years] | 24 [18 to 42]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Canada | 12

OUTCOME MEASURES:

1. Primary Outcome: Biodistribution of the 123I-CMICE-013 Within the Lungs
Description: SPECT imaging was performed immediately following 123I-CMICE-013 injection, after 90 min, 4 hours, 6 hours and 24 hours. Region of interest was manually drawn on planar images. The total number of counts in the full body region of interest of the initial images was taken to correspond to 100% of the injected dose. The uptake in the organ as a percentage to injected dose was calculated.
Time Frame: From enrollment to completion of imaging was 24 hours for each scan. Rest and stress scans were performed one week apart.
Population: Normal, healthy volunteers, with no pre-existing medical conditions were recruited. The volunteers were six (6) males and six (6) females and ranged from 18 to 42 years of age.
Measure: Mean (Standard Deviation); unit: percentage of total injected dose
Groups:
- Lung Biodistribution of 123I-CMICE-013 Post Rest Imaging; Lung Biodistribution of 123I-CMICE-013 Post Stress Imaging: Administration and analysis of alternative MPI radiotracer
  For SPECT imaging at rest, patients were injected with a 190 +/- MBq dose of 123I-CMICE-013 injected as a single bolus over 10-20 sec followed by a saline flush. Patients underwent SPECT imaging immediately following injection, after 90 in, 4 hours, 6 hours, and 24 hours. Regions of interest were manually drawn on planar images. The biodistribution of the 123I-CMICE-013 at rest was calculated.
Arm/Group | Lung Biodistribution of 123I-CMICE-013 Post Rest Imaging | Lung Biodistribution of 123I-CMICE-013 Post Stress Imaging
Number analyzed (Participants) | 12 | 12
percentage of total injected dose
  Biodistribution immediately after 123I-CMICE-013 injection. | 8.4 (1.9) | 7.1 (1.1)
  Biodistribution at 90 min post 123I-CMICE-013 injection | 7.1 (1.8) | 6.2 (1.0)
  Biodistribution at 4 hours post 123I-CMICE-013 injection | 5.3 (1.4) | 4.8 (0.9)
  Biodistribution at 6 hours post 123I-CMICE-013 injection | 4.3 (1.1) | 4.1 (0.8)
  Biodistribution at 24 hours post 123I-CMICE-013 injection | 0.8 (0.2) | 1.0 (0.2)

2. Primary Outcome: Biodistribution of the 123I-CMICE-013 Within the Thyroid
Description: as for outcome 1
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of total injected dose
Groups:
- Thyroid Biodistribution of 123I-CMICE-013 Post Rest Imaging; Thyroid Biodistribution of 123I-CMICE-013 Post Stress Imaging: Administration and analysis of alternative MPI radiotracer
  For SPECT imaging at rest, patients were injected with a 190 +/- MBq dose of 123I-CMICE-013 injected as a single bolus over 10-20 sec followed by a saline flush. Patients underwent SPECT imaging immediately following injection, after 90 in, 4 hours, 6 hours, and 24 hours. Regions of interest were manually drawn on planar images. The biodistribution of the 123I-CMICE-013 at rest was calculated.
Arm/Group | Thyroid Biodistribution of 123I-CMICE-013 Post Rest Imaging | Thyroid Biodistribution of 123I-CMICE-013 Post Stress Imaging
Number analyzed (Participants) | 12 | 12
percentage of total injected dose
  Biodistribution of 123I-CMICE-013 Immediately after injection | 0.8 (0.2) | 0.5 (0.1)
  Biodistribution 90 min post 123I-CMICE-013 injection | 0.7 (0.3) | 0.5 (0.1)
  Biodistribution 4 hours post 123I-CMICE-013 injection | 0.6 (0.3) | 0.4 (0.1)
  Biodistribution 6 hours post 123I-CMICE-013 injection | 0.5 (0.3) | 0.3 (0.1)
  Biodistribution 24 hours post 123I-CMICE-013 injection | 0.1 (0.1) | 0.1 (0)

3. Primary Outcome: Biodistribution of the 123I-CMICE-013 Within the Heart Wall
Description: SPECT imaging was performed at rest and at stress with each SPECT scan performed one week apart. SPECT imaging was performed immediately following 123I-CMICE-013 injection, after 90 min, 4 hours, 6 hours and 24 hours. Region of interest was manually drawn on planar images. The total number of counts in the full body region of interest of the initial images was taken to correspond to 100% of the injected dose. The uptake in the organ as a percentage to injected dose was calculated.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of total injected dose
Groups:
- Heart Wall Biodistribution of 123I-CMICE-013 Post Rest Imaging; Heart Wall Biodistribution of 123I-CMICE-013 Post Stress Imaging: Administration and analysis of alternative MPI radiotracer
  For SPECT imaging at rest, patients were injected with a 190 +/- MBq dose of 123I-CMICE-013 injected as a single bolus over 10-20 sec followed by a saline flush. Patients underwent SPECT imaging immediately following injection, after 90 in, 4 hours, 6 hours, and 24 hours. Regions of interest were manually drawn on planar images. The biodistribution of the 123I-CMICE-013 at rest was calculated.
Arm/Group | Heart Wall Biodistribution of 123I-CMICE-013 Post Rest Imaging | Heart Wall Biodistribution of 123I-CMICE-013 Post Stress Imaging
Number analyzed (Participants) | 12 | 12
percentage of total injected dose
  Biodistribution of 123I-CMICE-013 Immediately after injection | 5.0 (0.6) | 3.2 (0.6)
  Biodistribution after 90 min post 123I-CMICE-013 injection | 4.0 (0.4) | 2.6 (0.5)
  Biodistribution after 4 hours post 123I-CMICE-013 injection | 2.7 (0.3) | 2.0 (0.4)
  Biodistribution after 6 hours post 123I-CMICE-013 injection | 2.1 (0.3) | 1.6 (0.3)
  Biodistribution after 24 hours post 123I-CMICE-013 injection | 0.3 (0.1) | 0.4 (0.1)

4. Primary Outcome: Biodistribution of the 123I-CMICE-013 Within the Bladder
Description: as for outcome 1
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of total injected dose
Groups:
- Bladder Biodistribution of 123I-CMICE-013 Post Rest Imaging; Bladder Biodistribution of 123I-CMICE-013 Post Stress Imaging: Administration and analysis of alternative MPI radiotracer
  For SPECT imaging at rest, patients were injected with a 190 +/- MBq dose of 123I-CMICE-013 injected as a single bolus over 10-20 sec followed by a saline flush. Patients underwent SPECT imaging immediately following injection, after 90 in, 4 hours, 6 hours, and 24 hours. Regions of interest were manually drawn on planar images. The biodistribution of the 123I-CMICE-013 at rest was calculated.
Arm/Group | Bladder Biodistribution of 123I-CMICE-013 Post Rest Imaging | Bladder Biodistribution of 123I-CMICE-013 Post Stress Imaging
Number analyzed (Participants) | 12 | 12
percentage of total injected dose
  Biodistribution of 123I-CMICE-013 Immediately after injection | 3.6 (0.6) | 2.3 (0.6)
  Biodistribution 90 min post 123I-CMICE-013 injection | 5.3 (1.9) | 4.7 (1.8)
  Biodistribution 4 hours post 123I-CMICE-013 injection | 6.9 (3.9) | 4.8 (2.8)
  Biodistribution 6 hours post 123I-CMICE-013 injection | 6.0 (4.4) | 4.8 (2.8)
  Biodistribution 24 hours post 123I-CMICE-013 injection | 0.8 (0.3) | 1.0 (0.4)

5. Primary Outcome: Biodistribution of the 123I-CMICE-013 Within the Liver
Description: as for outcome 1
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of total injected dose
Groups:
- Liver Biodistribution of 123I-CMICE-013 Post Rest Imaging; Liver Biodistribution of 123I-CMICE-013 Post Stress Imaging: Administration and analysis of alternative MPI radiotracer
  For SPECT imaging at rest, patients were injected with a 190 +/- MBq dose of 123I-CMICE-013 injected as a single bolus over 10-20 sec followed by a saline flush. Patients underwent SPECT imaging immediately following injection, after 90 in, 4 hours, 6 hours, and 24 hours. Regions of interest were manually drawn on planar images. The biodistribution of the 123I-CMICE-013 at rest was calculated.
Arm/Group | Liver Biodistribution of 123I-CMICE-013 Post Rest Imaging | Liver Biodistribution of 123I-CMICE-013 Post Stress Imaging
Number analyzed (Participants) | 12 | 12
percentage of total injected dose
  Biodistribution of 123I-CMICE-013 Immediately after injection | 14.4 (2.1) | 9.0 (1.2)
  Biodistribution 90 min post 123I-CMICE-013 injection | 8.4 (0.9) | 5.9 (0.9)
  Biodistribution 4 hours post 123I-CMICE-013 injection | 5.4 (0.9) | 4.3 (0.9)
  Biodistribution 6 hours post 123I-CMICE-013 injection | 4.2 (1.0) | 3.7 (0.9)
  Biodistribution 24 hours post 123I-CMICE-013 injection | 0.7 (0.2) | 0.8 (0.2)

6. Secondary Outcome: Total Effective Dose of 123I-CMICE-013 for Men
Description: The uptake of 123I-CMICE-013 in each organ from the primary outcomes were used to calculate the dose to each organ using the Olinda/EXM software package. doses for male patients were calculated using the adult male model. The results are reported as the mean and standard deviation of those measurements over all male participants for both the rest and stress SPECT imaging scans.
Time Frame: as for outcome 1
Population: Normal, healthy volunteers, with no pre-existing medical conditions were recruited. The volunteers were six (6) males and ranged from 18 to 42 years of age.
Measure: Mean (Standard Deviation); unit: microsieverts per megabecquerel
Groups:
- Total Effective Dose of 123I-CMICE-013 for Men: For SPECT imaging at rest, patients were injected with a 190 +/- MBq dose of 123I-CMICE-013 injected as a single bolus over 10-20 sec followed by a saline flush. Patients underwent SPECT imaging immediately following injection, after 90 in, 4 hours, 6 hours, and 24 hours. The uptake of 123I-CMICE-013 in each organ from the primary outcomes were used to calculate the dose to each organ using the Olinda/EXM software package. doses for male patients were calculated using the adult male model. The results are reported as the mean and standard deviation of those measurements over all male participants for both the rest and stress SPECT imaging scans.
Arm/Group | Total Effective Dose of 123I-CMICE-013 for Men
Number analyzed (Participants) | 6
microsieverts per megabecquerel
  Total Effective Dose of 123I-CMICE-013 during Rest Imaging | 24.0 (5.0)
  Total Effective Dose of 123I-CMICE-013 during Stress Imaging | 23.0 (4.0)

7. Secondary Outcome: Total Effective Dose of 123I-CMICE-013 for Women
Description: The uptake of 123I-CMICE-013 in each organ from the primary outcomes were used to calculate the dose to each organ using the Olinda/EXM software package. doses for male patients were calculated using the adult female model. The results are reported as the mean and standard deviation of those measurements over all female participants for both the rest and stress SPECT imaging scans.
Time Frame: as for outcome 1
Population: Normal, healthy volunteers, with no pre-existing medical conditions were recruited. The volunteers were six (6) females and ranged from 18 to 42 years of age.
Measure: Mean (Standard Deviation); unit: microsieverts per megabecquerel
Groups:
- Total Effective Dose of 123I-CMICE-013 for Women: For SPECT imaging at rest, patients were injected with a 190 +/- MBq dose of 123I-CMICE-013 injected as a single bolus over 10-20 sec followed by a saline flush. Patients underwent SPECT imaging immediately following injection, after 90 in, 4 hours, 6 hours, and 24 hours. The uptake of 123I-CMICE-013 in each organ from the primary outcomes were used to calculate the dose to each organ using the Olinda/EXM software package. doses for female patients were calculated using the adult female model. The results are reported as the mean and standard deviation of those measurements over all female participants for both the rest and stress SPECT imaging scans.
Arm/Group | Total Effective Dose of 123I-CMICE-013 for Women
Number analyzed (Participants) | 6
microsieverts per megabecquerel
  Total Effective Dose of 123I-CMICE-013 during Rest Imaging | 30.0 (2.0)
  Total Effective Dose of 123I-CMICE-013 during stress Imaging | 29.0 (2.0)

ADVERSE EVENTS:
Groups:
- 123I-CMICE-013 Rest Dose: One resting dose of 185MBq administered on Day 1 of study participation.
- 123I-CMICE-013 Stress Dose: One stress dose of 185MBq administered on Day 8 of study participation.
Arm/Group | 123I-CMICE-013 Rest Dose | 123I-CMICE-013 Stress Dose
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 2/12 | 2/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 123I-CMICE-013 Rest Dose (N=12) | 123I-CMICE-013 Stress Dose (N=12)
Leg Injury (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — participant injured leg while undergoing scan
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) — Patient became nauseated during the scan
skin irritation (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Skin became irritated around injection site
Pressure spot (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — pressure spot on buttocks after scan completed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No